CLINICAL TRIAL: NCT01692639
Title: Acute Acetaminophen Ingestion: Does Repeated Acetaminophen Blood Test Have an Interest?
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5313
Record Dates: First submitted 2012-09-19; First posted 2012-09-25 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Acetaminophen Overdose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acetaminophen is the first drug involved in voluntary drug poisoning. According to the studies conducted in the USA and in the United Kingdom, it is the first cause of acute liver failure, and this poisoning is responsible of 10 percent of liver transplants each year in these countries. Mortality is about 1/3 at the stage of acute liver failure. The main risk factors are malnutrition and chronic alcoholism. Ease of access to this toxic and highly correlated with factors predisposing socio-economic field are an important issue, including the speed and appropriateness of care are key factors both in terms of reducing morbidity mortality in socio-economic terms for the community.A nomogram defines a statistical threshold from which the blood concentration of paracetamol has a significant risk of liver toxicity. The blood paracetamol dosage practiced today at the 4th hour after ingestion of a toxic dose, but there is no consensus on whether or not to repeat this dosage during the treatment, as the first result is beyond the threshold or not.The administration of the antidote NAC (N-acetyl-cysteine) in proven cases of liver toxicity is also regulated by a protocol that can vary in different services.In the absence of clear guidelines, the question of the need for iterative dosages of paracetamol blood beyond the fourth hour post-ingestion if the initial paracetamol blood measurement is below the curve nomogram remains open.Is it possible to limit blood tests to a single assay paracétamolémie to H4 when it is below the curve, and thus enable the return home of the patient's somatic point of view (excluding psychiatric care when is voluntary drug intoxication), with consequences in terms of costs (hospital days) and duration of treatment?

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Having taken a single dose of acetaminophen
* With a supposed ingested dose over 4 grams

Exclusion Criteria:

* Patients treated with N-Acetyl
* Cysteine before their admissions in the participating units
* With repeted ingested doses
* Pregnant and nursing wifes
* Patients unable to give their consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years with acute paracetamol ingestion admitted in a group of 8 emergency departments of the region Alsace, France (Strasbourg Hautepierre and Nouvel Hôpital Civil, Haguenau, Saverne,Wissembourg, Colmar, Sélestat, Mulhouse) and with a single dose of paracetamol over 4 grams.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal BILBAULT, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (10):
- France (10):
  - Centre Hospitalier Gérontologique, Bischwiller
  - Service d'accueil des Urgences, Hôpitaux Civils de Colmar, Centre Hospitalier Louis Pasteur, Colmar
  - Service d'Accueil des Urgences, Centre Hospitalier de Haguenau, Haguenau
  - Service des Urgences, CH Emile Muller, Mulhouse
  - Service des Urgences, Centre Hospitalier de Sélestat, Sélestat
  - Service d'Accueil des Urgences, Nouvel Hôpital Civil, Strasbourg
  - Service de Réanimation Médicale, Nouvel Hôpital Civil, Strasbourg
  - Service de Réanimation Médicale, Hôpital de Hautepierre, Strasbourg
  - Service des Urgences, Hôpital de Hautepierre, Strasbourg
  - Service des Urgences, Centre Hospitalier Intercommunal de la Lauter, Wissembourg